CLINICAL TRIAL: NCT01768065
Title: Nasal Expiratory Positive Airway Pressure for the Treatment of Pediatric Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Ignacio Tapia, MD, Principal Investigator, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-008691
Record Dates: First submitted 2013-01-10; First posted 2013-01-15 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Organic Pediatric Obstructive Sleep Apnea
Keywords: NEPAP; CPAP; alternative; OSAS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal Expiratory Positive Airway Pressure Devices (Experimental): Nasal Expiratory Positive Airway Pressure Device
  Interventions: Device: Nasal Expiratory Positive Airway Pressure Device
- placebo sham (Sham Comparator): A sham device
  Interventions: Device: placebo sham

INTERVENTIONS:
Device: Nasal Expiratory Positive Airway Pressure Device — assigned to Nasal Expiratory Positive Airway Pressure arm
  Arms: Nasal Expiratory Positive Airway Pressure Devices
Device: placebo sham
  Arms: placebo sham

SUMMARY:
This study will evaluate effectiveness and adherence of the nasal expiratory positive airway pressure (NEPAP) device as an an alternate therapy for children with Obstructive Sleep Apnea Syndrome (OSAS). NEPAP is currently approved for use only in adults.

DETAILED DESCRIPTION:
The nasal expiratory positive airway pressure (NEPAP) device has been used to treat OSAS in adults. A disposable device is placed in each nostril at night and attached with adhesive. The device acts as a one-way valve, during inspiration the valve opens, with negligible resistance to flow. During expiration, the valve closes and airflow is directed through small air channels, increasing resistance. The increased resistance helps to maintain the upper airway pressure during the critical end-expiratory period when the upper airway has been found to be most narrow in the breaths preceding an apnea event. In contrast to Continuous Positive Airway Pressure (CPAP) which provides positive pressure during both inspiration and expiration, NEPAP creates pressure during expiration. NEPAP is a potential alternative therapy which is less cumbersome than CPAP and may increase adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 5-16 years (note: Due to the size of the devices, it is expected that most children will be at least 8 years old, but a few may be younger. Subjects will be evaluated in clinic to fit for size and habituate to the device)
2. OSAS (AHI > 5/hr)
3. Subject has had adenotonsillectomy or is not a candidate for adenotonsillectomy
4. Subject is non-adherent to CPAP or is seeking an alternative therapy
5. Tolerance of NEPAP device during a daytime session
6. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Severe developmental delay thought to involve a high risk of aspiration
2. Family does not understand English well enough to perform the standardized, validated questionnaires.
3. Age >16 years since results may be similar to adult studies in these older patients.
4. Severe breathing disorder (including respiratory muscle weakness, bullous lung disease, bypassed upper airway, pneumothorax, pneumomediastinum)
5. Severe heart disease (including heart failure)
6. An acute upper respiratory (including nasal, sinus or middle ear) inflammation or infection or perforation of the ear drum

Subjects that do not meet all of the enrollment criteria will not be enrolled. Any violations of these criteria will be reported in accordance with Institutional Review Board (IRB) Policies and Procedures.

Study members will not recruit females who are known to be pregnant. However, if a subject becomes pregnant during the study, we will continue to use the device. Pregnancy is not an exclusion criterion as positive airway pressure therapy does not harm the pregnant woman or fetus.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index | Approximately one week
  The apnea hypopnea index during polysomnography will be compared between the active device and the placebo nights

SECONDARY OUTCOMES:
Adherence using daily logs | One month
  Adherence with using devices will be determined by daily logs and collecting used devices

OTHER OUTCOMES:
Quality of life | One Month
  The Pediatric Quality of Life (PedsQL) score will be compared at baseline and after one month of device usage

CONTACTS AND LOCATIONS:
Overall Officials: Carole Marcus, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kureshi SA, Gallagher PR, McDonough JM, Cornaglia MA, Maggs J, Samuel J, Traylor J, Marcus CL. Pilot study of nasal expiratory positive airway pressure devices for the treatment of childhood obstructive sleep apnea syndrome. J Clin Sleep Med. 2014 Jun 15;10(6):663-9. doi: 10.5664/jcsm.3796. PMID 24932147